CLINICAL TRIAL: NCT06275295
Title: Application of Transbronchial Cryobiopsy in the Diagnosis of Progressive Pulmonary Fibrosis：a Multicenter Retrospective Study
Brief Title: A Retrospective Study of Transbronchial Cryobiopsy in the Diagnosis of Progressive Pulmonary Fibrosis
Status: Not yet recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Other Study IDs: ZRJY2021-BJ08-03-01-01
Record Dates: First submitted 2024-02-17; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Pulmonary Fibrosis; Transbronchial Cryobiopsy
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the diagnostic effectiveness, safety, and influencing factors of transbronchial cryobiopsy（TBLC） in progressive pulmonary fibrosis.

DETAILED DESCRIPTION:
The goal of this observational study is to learn about the diagnostic effectiveness, safety, and influencing factors of transbronchial cryobiopsy（TBLC） in progressive pulmonary fibrosis. The main question it aims to answer are: • The diagnostic rate of MDD1 or MDD2 based on TBLC. • The rate of hemorrhage, pneumothorax, acute ILD exacerbation and mortality. Participants' medical records will be collected by us.

ELIGIBILITY:
Inclusion Criteria:

Patients with PPF, ≥18 years of age, unclassified ILD, HRCT ≤3 months, forced vital capacity (FVC)≥50% predicted value, pulmonary carbon monoxide diffusion (DLCO)≥35% predicted value, echocardiography ≤12 months, estimated pulmonary systolic blood pressure ≤40 mmHg, Body mass index (BMI)≤35 kg/m2.

Exclusion Criteria:

Patients with platelet counts below 50,000e+9/L or International Normalized ratio of prothrombin time (INR) above 1.5 are not eligible for TBLC

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving TBLC for progressive pulmonary fibrosis
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2024-12-24 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic rate of MDD2 based on TBLC | December，31，2024
  the diagnostic rate of progressive pulmonary fibrosis after Transbronchial Cryobiopsy

SECONDARY OUTCOMES:
The diagnostic rate of MDD1 | December，31，2024
  the diagnostic rate of progressive pulmonary fibrosis before Transbronchial Cryobiopsy